CLINICAL TRIAL: NCT07385651
Title: Deceased Donor Kidney Storage at 10 Celsius Versus Conventional Storage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Traferox Technology Inc. (Unknown)
Responsible Party: Principal Investigator, Christian Crannell, Assistant Professor of Surgery, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 241113
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: End Stage Chronic Renal Failure; Chronic Kidney Disease (Stages 4 and 5); Kidney Transplantation Recipients
Keywords: kidney transplant recipients; delayed graft function; ischemia reperfusion injury; 10 Celsius kidney storage
MeSH Terms: conditions — Renal Insufficiency, Chronic; Delayed Graft Function; Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: If the donor kidney is coming from an organ procurement organization(s) (OPO) participating in the trial, the study organ coordinator will alert the on-site procurement team that the kidney is to be placed at 10˚C (the intervention arm).
  If the donor kidney is outside of a participating OPO these organs are automatically stored on ice (the control arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 10˚C deceased donor kidney storage (Experimental): Deceased donor kidneys from participating organ procurement organizations (OPO) will be procured per OPO routine clinical practice and then stored at 10˚C in dedicated temperature controlled coolers until transplant at Vanderbilt University Medical Center. Donor kidneys will be labeled with the anonymous United Network for Organ Sharing number. The transplant will then proceed per routine clinical practice and usual clinical pathways will be followed. Post operatively, study participants will have their urine collected 24 hours post operatively and analyzed. Routine clinical information will be abstracted from the electronic medical record and used for analysis.
  Interventions: Device: 10˚C deceased donor kidney storage using Traferox XPort
- Conventional (ice storage) deceased donor kidney storage (No Intervention): Deceased donor kidneys, not meeting eligibility for the intervention arm, that are accepted for transplant at Vanderbilt University Medical Center will be procured per routine clinical practice and stored conventionally on ice. Donor kidneys will be labeled with the anonymous United Network for Organ Sharing number. The transplant will proceed per routine clinical practice. Usual clinical pathways will be followed. Post operatively, study participants will have their urine collected 24 hours post operatively and analyzed. Routine clinical information will be abstracted from the electronic medical record and used for analysis.

INTERVENTIONS:
Device: 10˚C deceased donor kidney storage using Traferox XPort — Deceased donor kidneys will be stored using the Traferox XPort device to maintain an organ temperature of 10˚C during storage and transport until the time of transplant
  Arms: 10˚C deceased donor kidney storage

SUMMARY:
The goal of this clinical trial is to test how storage temperature of deceased donor kidneys affects kidney function after transplant in adult patients receiving a kidney transplant.

The main question it aims to answer is:

• Do patients that receive a kidney transplant stored at 10 °C have improved post-transplant kidney function? Researchers will compare patients who receive kidneys stored at 10 °C versus kidneys stored at 4°C (on ice, i.e. conventional storage) to see if kidneys stored at 10 °C have improved function.

Participants will:

* Be made aware of and consent to receive a kidney transplant that had been stored at 10 °C
* Have their urine collected 24 hours after surgery to be analyzed for research

DETAILED DESCRIPTION:
Kidney transplantation is a life-saving treatment for patients with end stage kidney disease, which affects nearly 800,000 patients in the United States. However, deceased donor kidney transplantation is often complicated by delayed graft function (DGF), conventionally defined as the recipient requiring hemodialysis within the first week after transplant. DGF is unfortunately common, occurring in 25% of all transplanted kidneys and portends worse long-term graft survival, higher rates of rejection, and increased recipient mortality. DGF commonly occurs because of ischemic reperfusion injury (IRI), a complex pattern of injury occurring at the time of organ procurement. IRI results from decreased cellular ATP, decreased function of the Na/K pump, mitochondrial destabilization, the generation of reactive oxygen species (ROS), apoptosis, complement and immune cell activation. Most commonly, kidneys and other deceased donor organs have been stored at 4˚C (ie on ice) to minimize cellular oxygen consumption and prevent IRI. However, preliminary data show that porcine kidneys are exposed to high levels of ROS at 4˚C due to decreased mitochondrial protective pathways associated with hypothermic conditions. Promising studies in other organ systems demonstrate reduced ROS when organs are stored at 10˚C instead of on ice. In lung transplant, porcine lungs stored at 10˚C vs ice show better physiologic metrics, decreased mitochondrial DNA release, less cell death, less lactate production, and less glucose consumption. Higher levels of protective mitochondrial metabolites were observed in lungs stored at 10°C than on ice. These metabolites promote the innate anti-oxidative system within mitochondria, protecting against ischemic injury. Clinically, human lung transplant shows favorable clinical outcomes with prolonged cold ischemia at 10˚C vs ice. Within kidney transplant, there have been no similar investigations of 10˚C storage compared to ice. We hypothesize that deceased donor kidney storage at 10˚C will be superior to ice. This study has the potential to transform deceased donor organ storage and establish a new standard of care by storing kidneys at 10˚C. Further, preserving kidney mitochondrial function and decreasing the rate of DGF, would allow transplant centers to accept more organs by lowering the clinical risk associated with organ acceptance, with an overall increase in organ utilization.

Methods Once an organ offer is made to VUMC and reviewed for suitability, the kidney transplant recipient will be contacted by one of our research key study personnel (KSP), trained as kidney transplant organ coordinators to review the organ offer per standard operating procedure. Once the patient has accepted the organ offer, the coordinator will review the study with the patient using the phone script for informed consent.

Organ storage groups: 10˚C vs. ice The study will test the difference between storage of donor kidneys at 10˚C (experimental) and ice storage (standard of care). The storage method used will be determined by the location of the donor kidney because of study logistics (see below).

If the donor kidney is coming from organ procurement organization(s) (OPO) participating in the trial, the study organ coordinator will alert the on-site procurement team that the kidney is to be placed at 10˚C. The organ coordinators have regular and frequent contact with the OPOs as part of the procurement and transplant process. If the donor kidney is outside of a participating OPO, no alert is required. These organs are automatically stored on ice.

All donor kidneys will be obtained per standard clinical practice by the local procurement surgeon. After collection, the kidneys will either a) be placed in a temperature controlled portable cooler and maintained at 10˚C or b) be stored on ice per standard of care procedures. Donor kidneys will be labeled with the anonymous United Network for Organ Sharing number and transported to VUMC.

The kidney transplant will proceed per routine clinical practice at VUMC regardless of storage conditions. Standard VUMC kidney transplant practices and clinical pathways will be followed for each study arm. Immunosuppression protocols will be followed and identical for each arm.

Post operatively, study participants will have their urine collected 24 hours post operatively and analyzed. Routine clinical information will be abstracted from the electronic medical record and used for analysis.

ELIGIBILITY:
Participant inclusion criteria

1. All adult single organ kidney transplant candidates on the waiting list at Vanderbilt University Medical Center (VUMC) will be eligible for enrollment.

Participant exclusion criteria

1. Kidney transplant candidates less than 18 years old
2. Kidney transplant candidates that decline consent
3. Transplant candidates listed for multi-organ transplant

Deceased donor organ inclusion criteria:

1. Donation after brain death or donation after circulatory death kidney donors, whose health care proxy has consented for donation and the possibility of research
2. Deceased donor kidneys that have been allocated to VUMC as a primary match offer prior to organ procurement will be eligible

Deceased donor organ exclusion criteria:

1. Donors whose health care proxy has declined consent for the possibility of research
2. Deceased donor kidneys that have been allocated to VUMC as a backup offer
3. Deceased donor kidneys that have been allocated to VUMC as a post procurement offer
4. Deceased donor kidneys that have already been placed on ice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Urine NGAL | Urine collected post operatively day one after kidney transplant
  Neutrophil gelatinase-associated lipocalin (NGAL), a urine biomarker for acute kidney injury that has been shown to be predictive of delayed kidney graft function. Urine will be collected after the kidney transplant, processed and stored with an anonymous ID.

SECONDARY OUTCOMES:
Delayed graft function | Within 7 days after kidney transplant
  Delayed graft function is defined as the patient requiring dialysis within 7 days after kidney transplant.
Post operative urine output | 24 hours after kidney transplant
  Total volume of urine output for the first 24 hours after the kidney transplant
Creatinine and estimated glomerular filtration rate trends | One month post operatively after kidney transplant
  Participants serum creatinine and estimated glomerular filtration rate trends will be abstracted from the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: W. Christian Crannell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
This study is committed to promoting transparency and reproducibility in research. Individual Participant Data (IPD) underlying the results reported in this study will be made available upon reasonable request. Requests for access to IPD will be considered on a case-by-case basis, contingent on the provision of a methodologically sound proposal and compliance with ethical guidelines. Data sharing will occur in accordance with applicable privacy regulations, informed consent from participants, and institutional policies. Researchers wishing to access the data should contact the corresponding author. De-identified participant data such as demographic information that was collected as part of the study will be available. Results will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026 through January 2028
Access Criteria: Other researchers will be able to email the primary investigator to request: de-identified participant data, results, and other study materials including the protocol and blank informed consent documents. No identifiable participant data will be released.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT07385651/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT07385651/ICF_001.pdf